CLINICAL TRIAL: NCT04930952
Title: Complications of Ethanol-amine Oleate Intralesional Sclerotherapy Injections of Maxillofacial Venous Malformations in Pediatric Patients
Brief Title: Complications of Ethanol-amine Oleate Intralesional Sclerotherapy
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Sarah Arafat, Assistant Lecturer, Suez Canal University
Other Study IDs: 157-2018
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Venous Malformation
Keywords: Maxillofacial; Pediatric; Venous Malformations; Ethanol-amine Oleate
MeSH Terms: interventions — Sclerotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ethanol-amine Oleate Sclerotherapy Injection — Intralesional Sclerotherapy Injection
  Other Names: Sclerotherapy

SUMMARY:
The aim of this study is to clarify complications of Ethanolamine Oleate intralesional injections of maxillofacial venous formations in pediatric patients

DETAILED DESCRIPTION:
Maxillofacial Venous malformations cause many functional and esthetic complications in children, intralesional sclerotherapy is the best choice of treatment; and Ethanol-amine Oleate has been the most commonly used sclerosing agent.

The aim of this study is to clarify complications of Ethanolamine Oleate intralesional injections of maxillofacial venous formations

ELIGIBILITY:
Inclusion Criteria: maxillofacial venous malformation

-

Exclusion Criteria:

1. Patients with lung, liver, or kidney diseases
2. Patients with Klippel-Trenaunay syndrome
3. Patients mental or physical disabilities

Max Age: 12 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients of age up to 12 years having maxillofacial venous malformations
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 12 months
  Complete Response - Marked Improvement - Moderate Improvement - No Response

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Arafat, MSc, Principal Investigator — Assistant Lecturer
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided